CLINICAL TRIAL: NCT03555006
Title: Tele-ultrasound Experimentation: Cooperation Protocol Between Electro-radiology Assistant and Remote Radiologist for the Realization of Some Exploration Indications by Ultrasound
Brief Title: Tele-ultrasound Experimentation: Cooperation Protocol Between Electro-radiology Assistant and Remote Radiologist
Acronym: TELECHO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: because of the health crisis, organizational constraints and the lack of medical and paramedical staff
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-04-CHRMT
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Tele-ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local vs remote group (Other): The examination will be interpreted by a department's radiologist and by a remote radiologist in blind of the first interpretation
  Interventions: Other: Dual ultrasound reading "local vs remote"
- Local vs local group (Other): The examination will be interpreted by two department's radiologists
  Interventions: Other: Dual ultrasound reading "local vs local"

INTERVENTIONS:
Other: Dual ultrasound reading "local vs remote" — The examination will be interpreted by a department's radiologist and by a remote radiologist in blind of the first interpretation and a posteriori by a third radiologist.
  Arms: Local vs remote group
Other: Dual ultrasound reading "local vs local" — The examination will be interpreted by two department's radiologists and a posteriori by a third radiologist.
  Arms: Local vs local group

SUMMARY:
This study tries to evaluate the non-inferiority quality and safety of ultrasound examinations realise by electro-radiology assistant with a remote radiologist compared to those realize by electro-radiology assistant with a referent radiologist on site.

DETAILED DESCRIPTION:
The number of requests for medical imaging examinations is clearly growing while there is an understaffing among the radiologists. The solution is the amelioration of information transmission technologies, for organize a territorial teleradiology in order to care duty. Currently, in the ultrasound field, the investigators can't realize image transfer because analyse and expertise are made during examination and only reading of fixed images can't be enough for the examination interpretation.

The most part of other developed countries recognize a paramedical job devoted to ultrasound. Tele-ultrasound is used in expert resort, for example during high-risk pregnancy.

A French society commercializes tele-ultrasound robots, arranged by a caregiver beside sick person and a tele-radiologist realize acquisition of information and images with remote commands from robot.

The CHR Metz-Thionville has a cooperation protocol between electro-radiology assistants and radiologists for the ultrasound practical, endorsed by Lorraine ARS and HAS (French health organizations) since 2012, and currently national impact.

This study purpose to evaluation the non-inferiority of agreement between two interpretations of the same ultrasound realize by an electro-radiology assistant on the one hand by two radiologists present in the radiology service and on the other hand, one radiologist in by the radiology service and one remote radiologist.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Who needs abdomino-pelvic ultrasound, except emergency cases
* With no substitutable examination

Exclusion Criteria:

* Pregnant and nursing women
* Patient in the incapacity to express his consent
* Unavailability of a remote radiologist or a second local radiologist during the examination realization
* Patient opposed to use data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Percentage of consistency between the reports | Day 1
  It will be evaluated in blind by a third radiologist with the RADPEER scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth PARIZEL, MD, Principal Investigator — CHR Metz Thionville
Locations (1):
- CHR Metz Thionville, Metz, France